CLINICAL TRIAL: NCT06522204
Title: Comparing the Gastric Emptying Times of Underweight and Healthy-weight School-aged Children After Preoperative Precise Fluid Intake
Brief Title: Comparing the Gastric Emptying Times of Underweight and Healthy-weight School-aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 09-2023/11
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Preoperative Fasting
Keywords: gastric empyting; gastric volume; ultrasonography

STUDY DESIGN:
Intervention Model Description: Pediatric patients will be divided into two groups as underweight and normal weight. Children under the % percentile will be considered as underweight.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup Underweight (Experimental): Experimental: Underweight pediatric patient Underweight children aged 6-14 years, under 5% percentile, fasted for the night before planned surgery.
  Interventions: Drug: %5 Dextrose
- Group Normal weight (Active Comparator): Active Comparator: Normal weight pediatric patient Normal weight children aged 6-14 years, between 5-85% percentile, fasted for the night before planned surgery.
  Interventions: Drug: %5 Dextrose

INTERVENTIONS:
Drug: %5 Dextrose — All the patients will receive oral 3mL/kg 5%Dextrose
  Other Names: Group U; Group N

SUMMARY:
In the recent literature, preoperative fasting times for pediatric patients are limited to one hour for clear fluids. Studies related to gastric emptying times mostly searched for normal-weight children. These studies have claimed that 3 mL/kg of clear liquid can be allowed up to 1 hour before surgery. There is a lack of interest in the gastric emptying time of underweight pediatric patients during the preoperative period. Recent studies suggest that underweight children may experience rapid gastric emptying. This trial compares the gastric volume and emptying time after ingesting 3 mL/kg clear fluid in underweight and normal-weight pediatric patients in the preoperative period.

DETAILED DESCRIPTION:
After receiving informed consent from the children and their families, the American Society of Anesthesiologists (ASA) 1-2 pediatric patients between 6 and 14 years who will be recruited for elective surgery will be included in this study. The children under the 5% percentile will be accepted as underweight. After, the basal gastric volume will be calculated with the help of Ultrasonography (USG). The children will receive oral 3 mL/kg 5% dextrose. USG evaluation will be made every 5 minutes until the gastric volume reaches the basal level. Children reaching basal gastric volume will be accepted as suitable for the surgery. This study compares the gastric volume and emptying time after ingesting 3 mL/kg clear fluid in underweight and average-weight pediatric patients in the pre-operative period.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical state I or II
* Age 6 to 14 years.
* Gender: both sexes.
* Scheduled for non-gastrointestinal Tract elective day-case surgery under general anesthesia.

Exclusion Criteria:

* Parent/caregiver refusal
* Ages < 6 or > 14 years old
* Children with gastroesophageal reflux disease
* Renal failure
* Diabetes mellitus
* Cerebral palsy patients
* Mental retardation
* Esophageal strictures, achalasia, or any intestinal disease that may impair gastric emptying.
* Gastrointestinal system surgery and neurosurgical patients
* Emergency surgery
* Violation of the prescribed fasting times
* Refusing to drink prescribed clear fluid

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time | 90 minute after Dextrose ingestion
  Time until the gastric volume reaches the baseline level again

SECONDARY OUTCOMES:
Antral cross-sectional area | Every 5 minute until the ACSA decreased to the baseline value (assessed up to 90 minute after Dextrose ingestion).
  Antral cross-Section Area (ACSA) (cm2) maximal anteroposterior diameter (D1) and longitudinal diameter (D2) will be measured with ultrasound and calculated with that mathematical formula:
  ACSA(cm2) = Π x D1 x D2 / 4

CONTACTS AND LOCATIONS:
Overall Officials: Rafet YARIMOGLU, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)